CLINICAL TRIAL: NCT02087969
Title: Effectiveness of Dry Needling to Decrease Trigger Point Size and Increase Soft Tissue Extensibility in the Triceps Surae Muscle as Measured Via Musculoskeletal Ultrasound
Brief Title: Triceps Surae Trigger Point Size and Muscle Extensibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00052299
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2015-03

CONDITIONS: Limited Dorsiflexion; Limited Ankle Range of Motion
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dry Needling (Experimental): Dry Needling to Triceps Surae
  Interventions: Procedure: Dry Needling
- Stretching (Experimental): Subjects will be given a home exercise program of stretches which are commonly prescribed to improve ankle dorsiflexion.
  Interventions: Procedure: Stretching

INTERVENTIONS:
Procedure: Dry Needling
  Arms: Dry Needling
Procedure: Stretching
  Arms: Stretching

SUMMARY:
The purpose of this study is to determine the effectiveness of dry needling in improving ankle range of motion and functional outcomes. There have been an increasing number of studies on dry needling as an intervention for pain but none thus far that have studied functional outcome measures of the ankle. The study will include healthy male subjects between the ages of 18-30 years old randomized in to 3 intervention groups of: dry needling of the triceps surae, triceps surae stretching only, dry needling and stretching. The subjects who receive dry needling as an intervention will have the trigger point identified and dry needling performed while under musculoskeletal ultrasound visualization. The subjects will undergo pre and post intervention testing including Lower Quarter Y-Balance test, passive ankle dorsiflexion, closed chain half kneeling dorsiflexion, standing dorsiflexion, deep squat, multisegmental flexion as well as Marx Activity Level Scale. There will be 3 days between the initial testing/intervention and follow up. These outcomes will be the primary variables of interest. Ultrasound, Y balance testing, self stretching, and range of motion measurements are safe and pose no risk to the subject. Dry Needling has been found to be very safe and effective in the hands of physical therapists with a calculated risk of adverse events to be less than 0.04%.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-30 Years Old
* No history of ankle surgery
* No current ankle injuries

Exclusion Criteria:

* hypothyroidism
* fibromyalgia
* connective tissue disorders
* chronic pain
* bleeding disorders including use of anti-coagulants
* vitamin D and B12 deficiencies
* active sites of cancer
* local or systemic infections
* local skin lesions, local lymphedema
* peripheral vascular disease including varicose veins
* compromised immune system
* needle phobia

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change of Ankle Dorsiflexion Range Of Motion | Baseline and 10 Minutes
  Ankle range of motion measures will be record before and immediately after the intervention.
Change in Ankle Dorsiflexion Range of Motion | Baseline and 3 Days
  Ankle dorsiflexion will again be measured at three days after the intervention to determine short term effectiveness of results.

SECONDARY OUTCOMES:
Change in Y-Balance Test for the Lower Quarter | Baseline and 20 Minutes
  Test of balance and functional performance of lower extremities.
Change in Y Balance Test for the Lower Quarter | Baseline and 3 Days
  Y Balance Test for the Lower Quarter will be assessed again at 3 days after the intervention to assess short term effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Cook, PhD, PT, Principal Investigator — Duke University
Locations (1):
- Duke Sports Medicine, Durham, North Carolina, United States